CLINICAL TRIAL: NCT01577121
Title: Evaluation of the Utility of Indomethacin as Support Treatment in Women With Preterm Labor With Intact Membranes and High Risk of Intraamniotic Inflammation
Brief Title: Evaluation of the Use of Indomethacin as Co-treatment in Women With Preterm Labor and High Risk of Intraamniotic Inflammation
Acronym: INDOGEST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sara Varea (Other)
Responsible Party: Sponsor-Investigator, Sara Varea, Clinical Research Manager, Fundacion Clinic per a la Recerca Biomédica
Organization: Fundacion Clinic per a la Recerca Biomédica (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: INDOGEST
Record Dates: First submitted 2012-04-10; First posted 2012-04-13 (Estimated); Last update posted 2014-10-21 (Estimated); Status verified 2014-10

CONDITIONS: Preterm Labor With Intact Membranes
Keywords: Preterm labor
MeSH Terms: conditions — Obstetric Labor, Premature | interventions — Indomethacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Drug: placebo
- indomethacin (Experimental): 50 mg/ 6 hours of indomethacin oral use
  Interventions: Drug: indomethacin

INTERVENTIONS:
Drug: indomethacin — 50 mg / 6 hours during 5 days
  Arms: indomethacin
Drug: placebo — 50 mg / 6 hours during 5 days
  Arms: placebo

SUMMARY:
To demonstrate if indomethacin associated to conventional treatment for preterm labor is useful to delay delivery and to improve neonatal morbimortality in women with preterm labor with high risk of intraamniotic inflammation

DETAILED DESCRIPTION:
Randomised patients would be assigned to receive indomethacin either placebo oral use(50 mg every 6 hours during 5 days) to evaluate the efficacy of indomethacin as complementary treatment to increase the gestational age at delivery in women admitted with preterm labor and intact membranes with high risk of intraamniotic inflammation, defined as a gestational age at admission less than 28.0 weeks or those women from 28-32.0 weeks with a sonographic cervical length less than 15 mm

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with preterm labor admitted to hospital and treated with tocolysis
* pregnant women less than 28.0 and those women from 28.0 to 32.0 with a sonographic cervical length < 15 mm
* single pregnancy
* normal amniotic fluid
* normal arterial ductus

Exclusion Criteria:

* Age below 18 years
* previous use of indomethacin in the index pregnancy
* chorioamnionitis, preterm prelabour rupture of membranes or those fetal or maternal pathologies which could be responsible of an iatrogenic preterm delivery.
* oligohydramnios
* allergy to NSAID
* previous history of gastrointestinal bleeding
* use of NSAID contraindicated
* not adherence to the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2012-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Gestational age at delivery | before than 42 weeks of gestation
  number of weeks and days at delivery

SECONDARY OUTCOMES:
proportion of patients with spontaneous preterm delivery before 34 weeks of gestation | at the end of study (maximum 1 year)
  the participants will be followed until delivery. The proportion of patiens with spontaneous preterm delivery before week 34 will be available at the end of the study, once the last patient delivers.
Incidence of adverse events | 1 year (end of study)
  adverse events will be registered
Latency from admission to delivery | between initial admission and delivery (before 42 weeks of gestation)
  Latency from admission to delivery will be calculated
IL-6 levels in amniotic fluid and umbilical cord blood | delivery (maximum 42 weeks of gestational age)
  the investigators will determine the level of IL-6 in different samples
Number of emergency visits | between initial admission and delivery (before 42 weeks of gestation)
  Number of visits to emergency area will be registered
Neonatal morbidity | at the end of the study (1 year)
  neonatal morbidity will be registered:
  * admission to Neonatal Intensive Care Unit (NICU)
  * number of days of NICU admission
  * respiratory distress syndrome
  * intraventricular haemorrage
  * early onset neonatal sepsis
  * necrotizing enterocolitis
  * late neonatal sepsis
  * neonatal death.
Neonatal death | at the end of the study (1 year)
  Neonatal deaths will be registered

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic of Barcelona- Maternity, Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Wilson A, Hodgetts-Morton VA, Marson EJ, Markland AD, Larkai E, Papadopoulou A, Coomarasamy A, Tobias A, Chou D, Oladapo OT, Price MJ, Morris K, Gallos ID. Tocolytics for delaying preterm birth: a network meta-analysis (0924). Cochrane Database Syst Rev. 2022 Aug 10;8(8):CD014978. doi: 10.1002/14651858.CD014978.pub2. PMID 35947046